CLINICAL TRIAL: NCT06472531
Title: A Phase I/IIa Study of PET/CT Imaging Using INR101 Injection in Healthy Male Subjects and Patients With Suspected Prostate Cancer
Brief Title: A Study of PET/CT Imaging Using INR101 Injection in Healthy Male Subjects and Patients With Suspected Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yunhe Pharmaceutical (Tianjin) Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: INR101-I/IIa-01
Record Dates: First submitted 2024-05-20; First posted 2024-06-25 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-05

CONDITIONS: Healthy Male Subjects; Suspected Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- phase I (Experimental): Experimental: INR101 PET/ CT
  Drug: INR101.
  Interventions: Drug: INR101
- phase II (Experimental): Experimental: INR101 PET/ CT
  Interventions:
  Drug: INR101
  Interventions: Drug: INR101

INTERVENTIONS:
Drug: INR101 — • 9±1 mCi of INR101 will be injected intravenously prior to perform the PET/CT
  Other Names: INR101 PET CT
  Arms: phase I
Drug: INR101 — * 9±1 mCi of INR101 will be injected intravenously prior to perform the PET/CT
  * 7±1 mCi of INR101 will be injected intravenously prior to perform the PET/CT
  Other Names: INR101 PET CT
  Arms: phase II

SUMMARY:
Phase I/II study in the management of Healthy Male Subjects and patients with suspected prostate cancer.

DETAILED DESCRIPTION:
A multi-center, prospective, open-label, randomized Phase I/II diagnostic study designed for the management of healthy male subjects and patients with suspected prostate cancer.

Phase I Study Objective: The primary goal is to assess the biodistribution, dosimetry, pharmacokinetic (PK) attributes, and safety profile of INR101 injections in healthy Chinese male subjects. The specific endpoints include evaluating the safety, Standardized Uptake Value (SUV), Accumulation (%ID), Retention Time, Absorbed Dose, Effective Dose, and PK parameters in whole blood, plasma, and urine following an intravenous administration of INR101.

Phase II Study Objective: This phase aims to determine the diagnostic efficacy of INR101 injection PET/CT scans in patients with suspected prostate cancers. The principal aim is to ascertain the optimal imaging conditions, which involve determining the best dose and timing of administration. This will be gauged based on the diagnostic performance metrics-sensitivity, specificity, and accuracy-of the INR101 injection PET/CT at different dosages and imaging intervals, using prostate biopsy pathology results as the reference standard.

ELIGIBILITY:
Phase 1 Inclusion Criteria:

1. Males aged ≥18 years old
2. Good health status or no major illness, judged by the investigator based on the following assessments: medical history, physical examination, vital signs, 12-lead electrocardiogram, laboratory tests that are normal or abnormal but not clinically significant
3. Agree to use contraceptive measures from the day of signing the informed consent form until 3 months after drug administration, to avoid sperm donation;
4. The subjects/legally authorized representative/guardian understands the purpose and procedures of the trial, and signs the informed consent form.

Phase 2 Inclusion Criteria:

1. Males aged ≥18 years
2. ECOG score of 0 or 1
3. Subjects who are planned to undergo prostate biopsy for pathological examination after clinical assessment, with no contraindications for biopsy
4. Routine blood tests, liver and kidney function, and coagulation function meet the corresponding conditions
5. Agree to use contraceptive measures from the date of signing the informed consent form to 3 months after medication administration, to avoid sperm donation
6. The subject/legal authorized representative/guardian understands the purpose and procedures of the trial and signs the informed consent form

Phase 1 Exclusion Criteria:

1. Subjects who cannot complete INR101 imaging according to the requirements
2. Subjects who cannot complete pharmacokinetics sample collection according to the requirements
3. Serum virology examination (Heptitis B surface antigen,Anti-Treponema pallidum antibody,HIV antibodies,Antibody to Hepatitis C Virus) is abnormal, which is judged by the researchers to have clinical significance
4. History of mental illness
5. History of past malignant tumors
6. History of past heart-related diseases
7. History of significant brain diseases in the past
8. Suffering from severe and/or poorly controlled and/or unstable diseases that the researcher judges may affect the study
9. History of bleeding or coagulation disorders
10. History of alcohol abuse or drug abuse/dependency
11. Known allergy to the active ingredients of INR101 or its components
12. Participated in other clinical trials before screening or during screening, or plans to participate in other clinical trials during this study
13. The researcher judges that there are any medical diseases or other conditions that may affect safety, compliance or may affect the results of the study

Phase 2 Exclusion Criteria:

1. Subjects who are unable to complete the INR101 imaging as required
2. History of any other malignant tumors in the past
3. Subjects in other interventional clinical trials or subjects in clinical trials of radioactive therapeutic drugs before signing the informed consent form
4. Receiving any anti-tumor treatment before drug administration
5. Known allergy to the active ingredients of INR101 or its components Abnormal serum virology examination
6. Researchers judge that there are any medical diseases or other conditions that may affect safety, compliance or may affect the study results.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Phase I primary outcome: incidence of adverse events of INR101 injection | 7 days after administration
  Treatment-emergent adverse events (AEs) will be assessed and graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Phase I primary outcome:radiation dosimetry | 3 hours after administration
  Mean absorbed radiation doses were estimated using the source and target organ framework. Eight health subjects underwent serial INR 101 PET/CT scans at three time points following radiotracer injection: 5±5 min，30±5 min，60±10 min，120±10 min，180±20 min.
Phase I primary outcome:Tmax (Time to reach maximum plasma concentration) | 4 hours after administration
  Assessment of INR101 Tmax in whole blood 4 hours after administration
Phase I primary outcome:t1/2 (Elimination half-life) | 4 hours after administration
  Assessment of INR101 t1/2 in whole blood 4 hours after administration
Phase I primary outcome:AUC0-t (Area under the plasma concentration-time curve from time 0 to time t) | 4 hours after administration
  Assessment of INR101 AUC0-t in whole blood 4 hours after administration
Phase I primary outcome:AUC0-∞ (Area under the plasma concentration-time curve from time 0 to infinity) | 4 hours after administration
  Assessment of INR101 AUC0-∞ in whole blood 4 hours after administration
Phase I primary outcome:CL (Clearance) | 4 hours after administration
  Assessment of INR101 CL in whole blood 4 hours after administration
Phase I primary outcome:Cmax (Maximum plasma concentration) | 4 hours after administration
  Assessment of INR101 Cmax in whole blood 4 hours after administration
Phase I primary outcome:SUV-standardized uptake value | 3 hours after administration
  Assessment of INR101 uptake by PET scan by measuring standardized uptake value in the target organs.
Phase I primary outcome:%ID/g - percentage of injected dose per gram | 3 hours after administration
  Assessment of INR101 uptake by PET scan by measuring percentage of injected dose per gram of tissue in the target organs
Phase I primary outcome:residence time - residence time in the the target organs | 3 hours after administration
  Assessment of INR101 uptake by PET scan by measuring residence time in the target organs
Phase II primary outcome :diagnostic efficacy | 28 days after administration
  The sensitivity, specificity, and accuracy of INR101 PET/CT

SECONDARY OUTCOMES:
Phase II secondary outcome: Incidence of adverse events of INR101 injection | 7 days after administration
  Treatment-emergent adverse events (AEs) will be assessed and graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Zhang, Ph.D, Principal Investigator — The First Medical Center of the General Hospital of the Chinese People's Liberation Army; Jigang Yang, Ph.D, Principal Investigator — Beijing Friendship Hospital; Fugeng Liu, BD, Principal Investigator — Beijing Hospital; Xuejuan Wang, Ph.D, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Yunhe Pharmaceutical (Tianjin) Co., Ltd., Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No